CLINICAL TRIAL: NCT05950607
Title: Trial to Reduce Antimicrobial Use In Nursing Home Residents With Alzheimer's Disease and Other Dementias 2.0 (TRAIN-AD 2.0)
Brief Title: Trial to Reduce Antimicrobial Use in Nursing Home Residents With Alzheimer's Disease and Other Dementias 2.0
Acronym: TRAIN-AD 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: NIA R37AG032982
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Alzheimer Disease; Infections
MeSH Terms: conditions — Dementia; Alzheimer Disease; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAIN AD 2.0 (Experimental): Nursing homes randomized to the experimental arm will emply a multicomponent intervention among their providers designed to improve the management of suspected infections in residents with dementia. The components include: a.Orientation sessions for providers, b.On-line case based course for providers, c.Infection management algorithms for providers, d. Guidelines for providers to communicate with proxies, and e. Education booklet about infections in dementia for providers.
  Interventions: Behavioral: TRAIN AD 2.0
- Usual Care (Active Comparator): Nursing homes randomized to the conrol arm will employ usual care to manage nursing home residents with dementia with suspected infections.
  Interventions: Behavioral: TRAIN AD 2.0

INTERVENTIONS:
Behavioral: TRAIN AD 2.0 — The study intervention is a multi-component training program targeting direct care providers and healthcare proxies for NH residents with moderate to advanced dementia intended to improve the management of urinary tract infections (UTIs) and lower respiratory tract infections (LRIs). The components include: A. Provider Orientation: At NH start-up and q2 months providers will be offered orientations sessions involving two 15-minute presentations, one focused on the background and rationale for the program and one focused on describing the program components. B. A case-based on-line course, "Infection Management in Moderate to Advanced Dementia," C. Posters and pocket cards for providers displaying algorithms guiding appropriate antimicrobial initiation for suspected UTIs and LRIs that integrate patient preferences, and D. Proxies of ALL residents in the facility will be sent a booklet related to infection management for persons with moderate to advanced dementia. .

SUMMARY:
The goal of this pragmatic cluster randomized clinical trial is to compare management of suspected infection in nursing home residents with dementia The main questions it aims to answer whether residents with dementia in nursing homes randomized to use a multicomponent intervention to optimize suspected infection management ( versus usual care) use less antibiotics and fewer burdensome interventions.

DETAILED DESCRIPTION:
This 52-month study (8 months preparation; 34 months trial conduct; 10 months data analyses and manuscript preparation)is a parallel cluster ePCT of an intervention to improve infection management for suspected infections among residents with moderate to advanced dementia (N=600; N=300/arm) living in NHs (N=50; N=25/arm). Facilities are members of a provider managed care network, Iowa Health Care Quality Network ('Network'). The intervention will be similar to the original TRAIN-AD program, but adapted for moderate to advanced dementia and rolled out in the Network. At each intervention NH, the intervention will be implemented for 24-months. Control NHs will employ usual care. In all NHs, there will be a 2-month startup period, 12-month resident enrollment period, and 24-months data collection period (Figure 2). Eligible residents with dementia will be identified using the EHR and Minimum DataSet (MDS) and followed up to 12 months. Outcome data will be ascertained from the EHR. Randomization and program roll out will be at the facility level. Analyses at the resident level. Clinical outcomes compared between arms at 12 months will be: 1. Antimicrobial courses/person-year in residents with moderate to advanced dementia (primary outcome) and all residents with dementia (secondary outcome) (Aim 1); and 2. Number of burdensome procedures/person-year used to manage suspected infections among residents with moderate to advanced dementia and those at all stages of dementia including: hospital transfers, urine specimens, chest x-rays, and blood cultures (secondary outcomes) (Aim 2). A process evaluation of implementation will be conducted in the intervention arm based on the RE-AIM framework1 (Aim 3) using quantitative and qualitative data (stakeholder interviews).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60
2. A diagnosis of dementia (any type)
3. Cognitive Functional Scale (CFS) > 1
4. NH length of stay >90 days

The CFS score categorizes cognitive impairment status based on data in the electronic health record into: 1. None, 2. Mild, 3. Moderate, and 4. Severe (advanced). For the primary outcome, the analysis will be restricted to residents with a CFS score of 3 or 4.

Exclusion Criteria:

1. Less than 60 years of age
2. Living in nursing home for less than 90 days
3. Does not have diagnosis of dementia
4. Does not meet CFS >1 score

Ages: 60 Years to 106 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial use in residents with moderate to advanced dementia | 12 months
  Number of antimicrobial courses/person-year among residents with moderate to advanced dementia.

SECONDARY OUTCOMES:
Antimicrobial use in residents with dementia | 12 months
  Number of antimicrobial courses/person-year among residents with dementia at any stage.
Burdensome interventions in residents with moderate to advanced dementia | 12 months
  Number of burdensome interventions (hospital transfers, bladder catheterization, chest x-ray, blood cultures) used to evaluate suspected infections/person-year among residents withmoderate to advanced dementia.
Burdensome interventions in residents with dementia | 12 months
  Number of burdensome interventions (hospital transfers, bladder catheterization, chest x-ray, blood cultures) used to evaluate suspected infections/person-year among residents with dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mitchell, MD, MPH, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew SeniorLife, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No